CLINICAL TRIAL: NCT02266238
Title: Randomized Controlled Trial to Compare Therapeutic Effect of Digital Subtraction Angiography(DSA)，Ultrasound Guided Balloon Dilatation and Surgical Reconstruction in Arteria-venous Fistula(AVF) Stenosis in Maintenance Hemodialysis Patients
Brief Title: Stenosis of Arteria-Venous Fistula in Maintenance Hemodialysis Patients: Early Intervention Trial
Acronym: SAVEIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director, Division of Nephrology, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZHKI-HDVA-003
Record Dates: First submitted 2014-09-22; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Uremia; Arteriovenous Fistula; Stenosis
MeSH Terms: conditions — Uremia; Arteriovenous Fistula; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): DSA guided percutaneous balloon dilatation to expand the stenosis of arteriovenous fistula
  Interventions: Device: DSA guided percutaneous balloon dilatation
- Group 2 (Experimental): Ultrasound guided percutaneous balloon dilatation to expand the stenosis of arteriovenous fistula
  Interventions: Device: Ultrasound guided percutaneous balloon dilatation
- Group 3 (Experimental): Surgical reconstruction of the stenosis to reconstruction the lumen of arteriovenous fistula
  Interventions: Procedure: Surgical reconstruction

INTERVENTIONS:
Device: DSA guided percutaneous balloon dilatation — Under the guidance of DSA, balloon is introduced into the stenosis area, proper pressure is given to achieve balloon dilatation to expand the narrow AVF lumen.
  Arms: Group 1
Device: Ultrasound guided percutaneous balloon dilatation — Under the guidance of ultrasound, balloon is introduced into the stenosis area, proper pressure is given to achieve balloon dilatation to expand the narrow AVF lumen.
  Arms: Group 2
Procedure: Surgical reconstruction — Direct surgery to reconstruction the AVF lumen.
  Arms: Group 3

SUMMARY:
The purpose of this study is to compare the effect of DSA guided percutaneous balloon dilatation, ultrasound guided percutaneous balloon dilatation and surgical repair in the treatment of Stenosis of Arteria-Venous Fistula in Maintenance Hemodialysis Patients.

DETAILED DESCRIPTION:
Eligibility Criteria:

1. Patients with long-term maintenance hemodialysis with AVF as the vascular access;
2. Positive clinical examination signs of AVF stenosis （not all required） : (1) the visual examination: edema, prolonged bleeding time, hematoma, aneurysm or constriction of the fistula .(2) the palpation examination: a narrowing of the outflow vein or aneurysm formation. (3) the auscultation examination: high pitch and/or discontinuous murmur.
3. Doppler ultrasound /DSA/magnetic resonance angiography show the diameter of AVF fistula is >50% narrow than the adjacent segment of the fistula lumen.
4. Blood flow of the AVF is <500ml/min or monthly declines of the blood flow>25%.
5. Patient signed the informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with long-term maintenance hemodialysis with AVF as the vascular access;
2. Positive clinical examination signs of AVF stenosis （not all required） : (1) the visual examination: edema, prolonged bleeding time, hematoma, aneurysm or constriction of the fistula .(2) the palpation examination: a narrowing of the outflow vein or aneurysm formation. (3) the auscultation examination: high pitch and/or discontinuous murmur;
3. Doppler ultrasound /DSA/MRA show the diameter of AVF fistula is >50% narrow than the adjacent segment of the fistula lumen;
4. Blood flow of the AVF is <500ml/min or monthly declines of the blood flow>25%;
5. Patient signed the informed consent.

Exclusion Criteria:

1. allergic to the iodine contrast or gadolinium contrast agent;
2. local infection;
3. the presence of severe coagulation dysfunction (or long-term history of taking warfarin or ticlopidine);
4. the presence of severe artery steal syndrome;
5. stenosis of immature fistula or fistula <2 month after vascular anastomosis;
6. severe central venous stenosis;
7. discontinue hemodialysis treatment (such as to transfer to peritoneal dialysis or kidney transplant);
8. severe cardiac dysfunction (New York Heart Association cardiac functional classification III or worse), unstable angina pectoris, myocardial infarction, severe left ventricular hypertrophy, or severe vascular embolic disease;
9. participated in other clinical trials within 12 weeks;
10. alcohol and/or drug abusers, mental disorders;
11. patients not suitable as the subjects of this trial under the consideration of researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the patency rate of the AVF after intervention | 24 month
  the patency rate including the primary and the secondary patency rate

SECONDARY OUTCOMES:
The success rate of AVF stenosis interventions | 24 month
  Described as %.
The recurrence rate of AVF stenosis interventions | 24 month
  Described as %.
The side effects of AVF stenosis interventions | 24 month
  Described as %.Side effects including bleeding, infection, thrombosis, artery steal syndrome, heart failure, inadequate dialysis, etc.
The cost-effectiveness analysis of AVF stenosis interventions | 24 month
  Described as $.

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China